CLINICAL TRIAL: NCT01655043
Title: Absolute Quantification of Coronary Flow Reserve by Stress Perfusion MRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Principal Investigator, James Carr, director of cardiovascular imaging, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: STU00050900; 000598 (Other Grant/Funding Number: Astellas Pharma Global Development, Inc)
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Myocardial Ischemia
Keywords: Magnetic Resonance Imaging; regadenoson
MeSH Terms: conditions — Myocardial Ischemia | interventions — regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- coronary artery disease patients (Experimental): Patients with suspected coronary artery disease prospectively recruited for myocardial perfusion MRI. All subjects to receive 5 ml IV gadofoveset trisodium contrast (Ablavar, Lantheus) at both stress and rest. Stress to be induced using 5 ml intravenous (IV) regadenoson (Lexiscan, Astellas US LLC), and the effects of regadenoson were reversed with 50 mg IV aminophylline following the completion of stress imaging.
  Interventions: Drug: Regadenoson; Drug: gadofoveset trisodium

INTERVENTIONS:
Drug: Regadenoson — Regadenoson will be infused intravenously 0.4 mg/5 mL (0.08 mg/mL) as a single bolus.
  Other Names: Lexiscan
Drug: gadofoveset trisodium — All subjects to receive 5 ml IV gadofoveset trisodium contrast (Ablavar) at both stress and rest.
  Other Names: Ablavar

SUMMARY:
Coronary artery disease (CAD, coronary heart disease) is the leading cause of death in the U.S., causing 1 in 5 deaths in 2005. The current method for diagnosing coronary artery disease that is considered most accurate is coronary angiography however it involves risk and radiation. Alternatively nuclear imaging test and MRI stress test only permits the semi qualitative analysis of the myocardial perfusion images.

In this proposal the investigators will develop a means to calculate Coronary Flow Reserve (CFR) using the MRI. the investigators approach has the potential to reduce mortality from myocardial infarction by effecting a change in the patient management paradigm. Absolute quantification of myocardial perfusion will detect coronary stenosis and CAD in patients with more accuracy than the semi-quantitative or qualitative analysis of perfusion images. Measurement of Coronary Flow Reserve is important for the following reasons: decrease of coronary flow reserve has been identified as a first effect of CAD; it provides an objective measure of treatment efficacy.

The purpose of this study is to compare images from nuclear stress test and/or coronary angiography with Magnetic Resonance Imaging (MRI) that will evaluate subjects with coronary artery disease calculating myocardial blood flow using a novel MRI technique combined to an extracellular Gadolinium-based contrast agent and stressor agent

DETAILED DESCRIPTION:
The main hypothesis the investigators will test is that changes in myocardial blood volume, under physiologic stress, correlate with myocardial flow reserve as measured in low spatial resolution nuclear SPECT scans. Secondary hypothesis is that stress perfusion as quantified with bolus height corrected gadofosveset trisodium images, better correlate with SPECT perfusion than uncorrected, relative perfusion values.

The investigators propose implementing the scan protocol using a 1.5T or 3.0T MRI scanner. The investigators will scan a series of 20 patients recruited from the nuclear stress lab at Northwestern Memorial Hospital. These subjects will be approached and enrolled into a HIPPA Compliant, IRB approved research study to assess the effectiveness of myocardial perfusion and blood volume images to measure myocardial blood volume. Subjects will be scanned with a modified version of the clinical stress-perfusion protocol. Correlation analysis will be used to test the hypothesis that quantitative blood volume is an indicator of myocardial flow reserve.

ELIGIBILITY:
Inclusion Criteria:

Under an Institutional Committee on Human Research board approved protocol, 20 patients with a suspected myocardial ischemic disease with positive stress nuclear medicine test laboratory will be recruited in this prospective study. All subjects will be screened for GFR within 24 hours before the exam. All patients must have a GFR > 30 mL/min/1.73m2 to be included in the study.

All subjects will be selected following the Nephrogenic Systemic Fibrosis (NSF) guidelines. All dialysis patients or end-stage renal disease patients with a creatinine clearance of < 30mL/min will not be selected for the study to avoid NSF.

Exclusion Criteria:

1. Age 18 to 89 years;
2. Known contraindication to MR imaging (such as pacemaker placement, magnetic implants, etc);
3. Claustrophobia;
4. Inability to perform an adequate breath-hold for imaging,
5. Inability to provide informed consent;
6. all subjects will be will be screened for GFR within 24 hours before the exam and subjects presenting with GFR < 60 ml/min will be excluded;
7. Pregnant and lactating women;
8. Patients with hypersensitivity to gadolinium contrast agents, metoprolol, adenosine, or nitroglycerin;

10) Contra indication for Regadenoson

1. 2nd- or 3rd-degree AV block (except in patients with a functioning artificial pacemaker)
2. Sinus node disease (except in patients with a functioning artificial pacemaker)
3. Unstable angina
4. Acute myocardial infarction
5. Known or suspected bronchoconstrictive or bronchospastic lung disease (e.g., asthma)
6. Hypersensitivity to adenosine
7. Caffeine within 12-24 hours
8. Theophylline and Dipyridamole products within 24 hours

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Carr, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Rosamond W, Flegal K, Friday G, Furie K, Go A, Greenlund K, Haase N, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell CJ, Roger V, Rumsfeld J, Sorlie P, Steinberger J, Thom T, Wasserthiel-Smoller S, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2007 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2007 Feb 6;115(5):e69-171. doi: 10.1161/CIRCULATIONAHA.106.179918. Epub 2006 Dec 28. No abstract available. PMID 17194875
- [Result] Elkington AG, Gatehouse PD, Ablitt NA, Yang GZ, Firmin DN, Pennell DJ. Interstudy reproducibility of quantitative perfusion cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2005;7(5):815-22. doi: 10.1080/10976640500287877. PMID 16353442
- [Result] Wu KC, Zerhouni EA, Judd RM, Lugo-Olivieri CH, Barouch LA, Schulman SP, Blumenthal RS, Lima JA. Prognostic significance of microvascular obstruction by magnetic resonance imaging in patients with acute myocardial infarction. Circulation. 1998 Mar 3;97(8):765-72. doi: 10.1161/01.cir.97.8.765. PMID 9498540

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Coronary Artery Disease Patients
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 20 participants with suspected coronary artery disease
Arm/Group | Coronary Artery Disease Patients
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Quantification of Myocardial Blood Volume
Description: The investigators anticipated that a novel MRI imaging protocol using a high relaxivity blood-pool contrast agent (gadofosveset trisodium) would be capable of quantifying coronary flow reserve based on quantification of myocardial blood volume and would be correlated with myocardial flow reserve as measured in low spatial resolution nuclear SPECT scans. Pre- and post- gadofosveset trisodium images were to be used to calculate the myocardial blood volume. Myocardial blood volume is derived from an equation of the relaxation times of hydrogen atoms in the blood and myocardium. If the agent administered did not behave as a true intravascular agent in the myocardium, quantification of myocardial intravascular blood volume (and hence a calculated coronary flow reserve) could not be calculated using the specified approach. In this case, relaxation times would be reported. Relaxation (R) times are measured in inverse seconds.
Time Frame: outcome measured following single MRI scan
Measure: Mean (Standard Deviation); unit: seconds^-1
Arm/Group | Coronary Artery Disease Patients
Number analyzed (Participants) | 20
seconds^-1
  Delta R1(blood) | 3.63 (.54)
  Delta R1(myo) | 1.23 (.24)

ADVERSE EVENTS:
Arm/Group | Coronary Artery Disease Patients
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
The small number of subjects results in reduced statistical power; The cohort was selected from patients at a single medical center, potentially reducing generalizability

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No